CLINICAL TRIAL: NCT00886717
Title: Open-label, Multicenter, Phase I/II Trial to Evaluate Efficacy Safety of the Combination Therapy of Genexol-PM and Carboplatin as a Firstline Treatment in Subjects With Advanced Ovarian Cancer
Brief Title: Paclitaxel-Loaded Polymeric Micelle and Carboplatin as First-Line Therapy in Treating Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: AMC-UUCM-GPMOC201; CDR0000639513 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-12

CONDITIONS: Ovarian Cancer
Keywords: stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage IIIA ovarian germ cell tumor; stage IIIB ovarian germ cell tumor; stage IIIC ovarian germ cell tumor; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; genexol-PM

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel-loaded polymeric micelle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel-loaded polymeric micelle and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of paclitaxel-loaded polymeric micelle and carboplatin and to see how well they work as first-line therapy in treating patients with advanced ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of paclitaxel-loaded polymeric micelle and carboplatin as first-line therapy in patients with advanced ovarian cancer. (Phase I)
* Evaluate the efficacy of this regimen, in terms of CA-125 response rate after 6 courses of therapy. (Phase II)

Secondary

* Assess, preliminarily, the antitumor activity of this regimen, in terms of objective response rate (complete response and partial response), time to tumor progression, and progression-free survival, in these patients. (Phase I)
* Evaluate the safety profiles of this regimen in these patients. (Phase I)
* Determine the objective response rate, as measured by RECIST criteria, in patients treated with this regimen. (Phase II)
* Determine the overall survival of patients treated with this regimen. (Phase II)
* Determine the overall response in patients treated with this regimen. (Phase II)
* Evaluate the safety and toxicity of this regimen in these patients. (Phase II)

OUTLINE: This is a multicenter study.

Patients receive paclitaxel-loaded polymeric micelle and carboplatin.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced ovarian cancer
* Measurable disease by RECIST criteria
* No prior or concurrent CNS metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 6 months
* Clinically acceptable blood, kidney, and spleen function
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No preexisting sensory or motor neuropathy ≥ grade 1
* No other malignancies within the past 5 years

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for ovarian cancer
* No prior immunotherapy or hormonal therapy for ovarian cancer
* No prior radiotherapy to the pelvis or abdominal cavity
* More than 2 weeks since prior major surgery other than debulking surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2008-05

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose (Phase I)
Efficacy, in terms of CA-125 response rate after 6 courses of therapy (Phase II)

SECONDARY OUTCOMES:
Preliminary antitumor activity, in terms of objective response rate (complete response and partial response), time to tumor progression, and progression-free survival (Phase I)
Safety profiles (Phase I)
Objective response rate as measured by RECIST criteria (Phase II)
Overall survival (Phase II)
Overall response (Phase II)
Safety and toxicity (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Man Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center at Yonsei University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center - University of Ulsan College of Medicine, Seoul